CLINICAL TRIAL: NCT00139126
Title: Research to Improve Smoke Alarm Functioning and Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Pacific Institute for Research and Evaluation (Other)
Responsible Party: Michael Ballesteros, CDC/NCIPC
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CDC-NCIPC-4662
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Wounds and Injuries; Burns
MeSH Terms: conditions — Wounds and Injuries; Burns

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Behavioral: Fire safety education — Education on smoke alarm maintenance based on behavioral theories

SUMMARY:
The purpose of this study to evaluate whether (1) targeted smoke alarm education, (2) general fire safety education with a smoke alarm component, (3) basic fire safety education, or (4) an unrelated intervention is most effective way to improve smoke alarm maintenance and function.

ELIGIBILITY:
Inclusion Criteria:

* live within four target neighborhoods in Prince George's County, MD that are at high risk for residential fire and injury.

Exclusion Criteria:

* primary decision maker of home is less than 18 years old
* speak a language other than english or spanish
* nobody at home after six return visits to the home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Actual)
Dates: Start 2005-08; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Smoke alarm functionality post-intervention. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Les R Becker, PhD, Study Director — Pacific Institute for Research and Evaluation; Ted R. Miller, PhD, Principal Investigator — Pacific Institute for Research and Evaluation
Locations (1):
- Pacific Institute for Research and Evaluation, Calverton, Maryland, United States

REFERENCES:
- [Derived] Miller TR, Bergen G, Ballesteros MF, Bhattacharya S, Gielen AC, Sheppard MS. Increasing smoke alarm operability through theory-based health education: a randomised trial. J Epidemiol Community Health. 2014 Dec;68(12):1168-74. doi: 10.1136/jech-2014-204182. Epub 2014 Aug 27. PMID 25165090